CLINICAL TRIAL: NCT07288671
Title: Effects of a Nostalgia Intervention on Alleviating Loneliness Amongst Community-dwelling Older Adults: A Cluster-randomised Waitlist-controlled Trial
Brief Title: Nostalgia Intervention on Alleviating Loneliness Amongst Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cho Lee Wong, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025.020-T
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Loneliness
Keywords: loneliness; older adults; nostalgia intervention

STUDY DESIGN:
Intervention Model Description: Wait-list trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Nostalgia intervention (Experimental): In addition to usual community support services, participants in the intervention group will receive the face-to-face nostalgia intervention weekly for 5 weeks (each session lasting approximately 90 minutes), with each group consisting of 5-8 older adults.
  Interventions: Behavioral: Nostalgia intervention
- Wait-list control (No Intervention): Participants in the wait-list control group will receive usual community support services provided by the community centres they belong to.

INTERVENTIONS:
Behavioral: Nostalgia intervention — Participants in the intervention group will receive the face-to-face nostalgia intervention weekly for 5 weeks (each session lasting approximately 90 minutes), with each group consisting of 5-8 older adults. The intervention consists of 5 sessions: Session 1 (understanding nostalgia and its benefits), Session 2-4 (music/ photos/ meaningful objects and nostalgia), Session 5 (reaffirming the benefits of nostalgia).
  Arms: Experimental: Nostalgia intervention

SUMMARY:
The proposed study will utilise a two-arm, cluster-randomised, waitlist-controlled trial to (1) examine the effects of the nostalgia intervention on loneliness, negative emotions, social connectedness, meaning in life and nostalgia amongst community-dwelling older adults in Hong Kong; (2) investigate whether the effect of the nostalgia intervention on loneliness is mediated by improvements in negative emotions, social connectedness and meaning in life; and (3) explore the experiences and perceptions of older adults participating in the nostalgia interventions, focusing on their views regarding the impact of the intervention on their loneliness.

DETAILED DESCRIPTION:
A convenience sample of 294 older adults from six participating community centres, with 49 participants from each centre. Eligible older adults will be randomly assigned to either a waitlist control group (n = 147) or an intervention group (n = 147). Both groups will receive standard community support services, whilst the intervention group will also participate in five weekly face-to-face nostalgia sessions (approximately 90 min each) in a group format. Additionally, a purposive subsample of 30 participants from the intervention group will be invited for focus group interviews.

The primary outcome (loneliness) and secondary outcomes will be assessed at baseline (T0), immediately post-intervention (T1), 3 months post-intervention (T2) and 6 months post-intervention (T3) using validated questionnaires. The investigators will analyse the quantitative data using a generalised estimating equation model with intention-to-treat and path analyses. The qualitative data will be analysed using reflexive thematic analysis. The findings of this proposed study will inform healthcare professionals and policymakers, offering practical strategies to combat loneliness in this vulnerable group.

ELIGIBILITY:
Inclusion Criteria:

* older adults aged 60 years or above
* residing in the community
* capable of speaking and understanding Chinese
* experiencing loneliness (scoring ≥3 on a three-item loneliness screening scale)

Exclusion Criteria:

* currently undergoing psychological intervention
* having a clinical diagnosis of mental illness
* being cognitively impaired (Abbreviated Mental Test score <6)
* having visual/language/communication difficulties

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Emotional and social loneliness | Asessed at baseline (T0), immediate after (T1), 3 months (T2), and 6 months (T3) post-intervention
  The Chinese version of the De Jong Gierveld Loneliness Scale. This six-item scale scores range from 0 to 6, with higher score indicates higher level of loneliness. This scale demonstrates good internal consistency (Cronbach's α = 0.76) and inter-rater reliability (ICC = 0.98-1.00), as well as a strong correlation with direct assessments of loneliness.
Existential Loneliness | Asessed at baseline (T0), immediate after (T1), 3 months (T2), and 6 months (T3) post-intervention
  Existential Loneliness Questionnaire, which comprises 22 items focused on loneliness in social ties, loneliness in close relationships and the search for meaning in life. The scores range from 22 to 132, higher scores indicate higher level of existential loneliness. The questionnaire also demonstrates good internal consistency (Cronbach's α = 0.90).

SECONDARY OUTCOMES:
Negative emotions | Asessed at baseline (T0), immediate after (T1), 3 months (T2), and 6 months (T3) post-intervention.
  The Chinese version of the Depression Anxiety Stress Scale consists of 21 items that assess symptoms of depression (7 items), anxiety (7 items), and stress (7 items). Each subscale scores range from 0 to 21, with higher scores indicating greater levels of negative emotions. The Chinese version demonstrates good internal consistency (Cronbach's α = 0.92 to 0.94).
Social connectedness | Asessed at baseline (T0), immediate after (T1), 3 months (T2), and 6 months (T3) post-intervention
  The revised Social Connectedness Scale to measure the perceived connection of participants to others in their social environment. This scale comprises 20 items measuring four aspects: belongingness, closeness, support and satisfaction. The scores range from 20 to 120, higher scores indicate greater feelings of social connectedness. This scale demonstrates good internal consistency (Cronbach's α = 0.92) and validity.
Meaning in life | Asessed at baseline (T0), immediate after (T1), 3 months (T2), and 6 months (T3) post-intervention.
  Meaning in Life Questionnaire, which comprises 10 items measuring presence for and search for meaning in life, to measure meaning in life. The score ranges from 10 to 70, higher scores indicates stronger sense of meaning in life. The Chinese version demonstrates good internal consistency (Cronbach's α = 0.85).
Nostalgia | Asessed at baseline (T0), immediate after (T1), 3 months (T2), and 6 months (T3) post-intervention
  The Southampton Nostalgia Scale to measure participants' nostalgia. This scale comprises five items that measure the importance participants attribute to nostalgia and two items related to frequency of nostalgia. The scores range from 7 to 49, higher scores indicate a greater dispositional tendency toward nostalgia. This scale demonstrates good internal consistency (Cronbach's α = 0.93).
Experiences and perceptions of older adults in intervention group | Assessed within 1 day (T1) after the intervention
  Focus group interviews will be conducted to explore the experiences and perceptions of older adults in intervention group regarding their participation in nostalgia interventions and the impact of the intervention on their loneliness using an interview guide.

CONTACTS AND LOCATIONS:
Overall Officials: Cho Lee Wong, PhD, Principal Investigator — The Nethersole School of Nursing, CUHK

IPD SHARING:
Plan to Share IPD: No